CLINICAL TRIAL: NCT02102919
Title: Skilling-up Exercise for Elderly in Need of Care
Brief Title: Innovative Training Program for Elderly in Need of Care Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Goethe University (Other); Maastricht University Medical Center (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Heiner Baur (PhD), PhD, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Main study (PhD)- part I
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Poor Performance Status; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): T0 - intervention over 4 weeks with stochastic resonance whole-body vibration (SR-WBV) (start with 3 up to 6 Hz, noise 4) T1 - intervention 4 weeks (SR-WBV (start with 3 up to 6Hz, noise 4 & virtual games) - T2
  Interventions: Device: SR-WBV; Device: Virtual Games (VG)
- Sham Comparator (Sham Comparator): T0 - intervention 4 weeks (SR-WBV 1 Hz, noise 1) - T1 - intervention 4 weeks (SR-WBV 1 Hz, noise 1 & Aktiv Tramp) - T2
  Interventions: Other: SR-WBV; Device: Aktiv Tramp (Swiss Frei AG, Switzerland)

INTERVENTIONS:
Device: SR-WBV — Participants will undergo a training program set over eight weeks, three times a week with 3 to 6 Hz, Noise 4.
  Other Names: SRT Zeptor® med
  Arms: Intervention group
Device: Virtual Games (VG) — Participants will undergo a training program set from week 5 to 8, three times a week over 20 minutes.
  Other Names: Virtual game board
  Arms: Intervention group
Other: SR-WBV — Participants will undergo a training program set over eight weeks three times a week with 1 Hz, Noise 1.
  Other Names: SRT Zeptor® med
  Arms: Sham Comparator
Device: Aktiv Tramp (Swiss Frei AG, Switzerland) — Participants will undergo a training program set from the 5 to 8 week, three times a week with 1Hz.
  Other Names: Mechanically controlled trampoline.
  Arms: Sham Comparator

SUMMARY:
The goal of this randomized controlled study was to examine the effects of a 8 weeks innovative training regime (stochastic resonance whole-body vibration [SR-WBV] and virtual virtual games [VG]) in the skilling up phase on physical performance and strength in elderly in need of care population.

DETAILED DESCRIPTION:
Sensorimotor and strength exercise are methods to increase strength & power in the field of geriatrics. The question that arise what exercises are best suited to and most effective for elderly in need of care individuals. Such populations are advised first to enter a "skilling up program" before more traditional forms of training exercises are implemented.

Goals in the skilling up phase: improvement in neuromuscular control, postural control and strengthening of large muscle groups of the lower extremity.

The aim of the study in the skilling up phase:

Study the effect on physical performance Study the effects on muscle strength.. The participants will be recruited in Canton Bern - Switzerland and will be randomly allocated to an intervention group or sham group.

ELIGIBILITY:
Inclusion Criteria:

* RAI (Resident Assessment Instrument) >0
* live in canton Bern
* in terms of training load be resistant.

Exclusion Criteria:

* acut joint disease, acut thrombosis, acute fractures, acute infections, acute tissue damage, or acute
* surgical scars
* seniors with prosthesis.
* alcoholic
* acute joint disease, activated osteoarthritis, rheumatoid arthritis, acute lower limb
* acute inflammation or infection tumors
* fresh surgical wounds
* severe migraine
* epilepsy acute severe pain

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Physical performance | after 8 weeks
  Short physical performance battery (SPBB): The SPBB examines 3 areas of lower extremity function: standing balance (semi-tandem stand, side-by-side stand, full tandem stand), usual walking speed and ability to stand from a chair. These areas represent essential tasks important for independent living.

SECONDARY OUTCOMES:
Isometric maximum voluntary contraction (IMVC) | after 8 weeks
  It will be evaluated by isometric MCV at 90 degree angle in the knee joint.
Submaximal maximum voluntary contraction (subIMVC) | after 8 weeks
  It will be evaluated by isometric RFD at 90 degree angle in the knee joint.
Isometric rate of force development (IRFD) | after 8 weeks
  It will be evaluated by isometric RFD at 90 degree angle in the knee joint.

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Baur, PhD, Principal Investigator — BUAS; Lorenz Radlinger, PhD, Study Director — Bern University of Applied Science, Department WGS; Eling Douwe de Bruin, PhD, Study Director — Swiss Federal Institute of Technology; Rob de Bie, Prof., Study Director — Maastricht University Medical Center; Dietmar Schmidtbleicher, Prof, Study Director — Goethe University
Locations (1):
- Slavko Rogan, Bern, Switzerland

REFERENCES:
- [Result] Rogan S, Radlinger L, Baur H, Schmidtbleicher D, de Bie RA, de Bruin ED. Sensory-motor training targeting motor dysfunction and muscle weakness in long-term care elderly combined with motivational strategies: a single blind randomized controlled study. Eur Rev Aging Phys Act. 2016 May 28;13:4. doi: 10.1186/s11556-016-0164-0. eCollection 2016. PMID 27239241